CLINICAL TRIAL: NCT03978741
Title: Randomized, Comparator-controlled, Single Blinded, Multi-center Study Evaluating the Efficacy and Safety of Yoni.Fit in Women With Stress Urinary Incontinence
Brief Title: Study Evaluating the Efficacy and Safety of Yoni.Fit in Women With Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Watkins Conti Products. Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-02041
Record Dates: First submitted 2019-05-08; First posted 2019-06-07 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Test Device (Experimental): Yōni.Fit Test Device
  Interventions: Device: Yōni.Fit Test Device
- Comparator Device (Active Comparator): Yōni.Fit Comparator Device
  Interventions: Device: Yōni.Fit Comparator Device

INTERVENTIONS:
Device: Yōni.Fit Test Device — The Yōni.Fit Test Device is a silicone pessary.
  Arms: Test Device
Device: Yōni.Fit Comparator Device — The Yōni.Fit Comparator Device is a silicone pessary with a different configuration.
  Arms: Comparator Device

SUMMARY:
Study to evaluate the safety and effectiveness of Yoni.Fit for the temporary management of stress urinary incontinence (SUI) in women.

DETAILED DESCRIPTION:
Randomized, comparator-controlled, single blinded, multicenter study to demonstrate the effectiveness, user acceptance, safety and tolerability of Yoni.Fit in the temporary management of stress urinary incontinence (SUI) in women.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be female,
2. Must be 18 years of age or older at the time of signing the informed consent
3. With BMI < 35
4. Must meet the following 2 criteria for diagnosis of stress urinary incontinence (SUI) :

   1. SUI clinical diagnosis via the cough supine test, AND
   2. ≥ 3 month history of experiencing Stress Urinary Incontinence (SUI) symptoms per the patient
5. Women of childbearing potential not intending to become pregnant for the duration of study participation. Subject must agree for the duration of the study to use one of the following forms of contraception

   1. Systemic hormonal treatment including oral pills, patches and injections OR
   2. "Single-barrier" contraception (condom, diaphragm and spermicide are each considered a barrier) OR
   3. Essure® procedure done at least three month prior to screening
6. Willing to comply with study requirements, including capable of performing the activities required for the pad weight test and return for follow-up visits.
7. Must be able to speak, understand and read English and sign study specific Informed Consent Form

Exclusion Criteria:

1. Women having predominantly urge or mixed incontinence as defined by:

   1. QUID Urge score >6, OR
   2. MESA percentage Urge Score > MESA percentage Stress Score Note: the questionnaires above will be self-administered and results interpreted by the subjects as per instructions in the questionnaires.
2. Current pregnancy, lactation or planning for pregnancy in the next 6 months
3. Women at postpartum for 3 months or less prior to screening
4. Women currently have an intrauterine device (IUD) as a contraception method placement less than 6 months or have an IUD over 6 month but may replace it next 14 weeks
5. Women currently use, have used an intra-vaginal device as contraception method for the past 6 months
6. Women currently using a pessary or treated previously with any device for UI
7. Women who have been treated with pharmacologic medications for UI within the past 4 months prior to screening, including any antidiuretic or diuretic medications (both over the counter and prescription medications)
8. Women who have been previously treated with any surgical or electrical interventions for UI
9. Women who have been previously treated with pelvic floor muscle training (PFMT) for UI within the past 4 months prior to screening
10. Women who have difficulty inserting or wearing an intra-vaginal device, including a tampon
11. Women who participated in a clinical trial within the 12 months prior to screening
12. Any of the following known conditions deemed prohibitory:

    1. Abnormal kidney function, including kidney stone
    2. Abnormal post void residual (e.g. greater than 150cc) or self-reported difficulty emptying bladder
    3. Allergy to silicon products and materials
    4. Acute febrile illness of any cause in the 14 days prior to screening
    5. Bladder stones or Bladder tumors
    6. Chronic pelvic pain within the past 4 months prior to screening
    7. Coagulation abnormalities
    8. Experience pain or burning sensation during sexual intercourse or urination
    9. Infections of the vagina, bladder and/or urethra within previous 3 months such as urinary tract infection (UTI)
    10. Interstitial cystitis
    11. Neurological disorders such as multiple sclerosis, spina bifida, Parkinson's disease which may interfere with nerve function of the bladder.
    12. Toxic shock syndrome (TSS) history or symptoms consistent with TSS
    13. Uncontrolled diabetes
    14. Undiagnosed vaginal bleeding or hematuria
    15. Vaginal discharge with a strong odor and irritation within previous 3 months
    16. Vaginal soreness or pain or fibromyalgia or paravaginal defect
13. Any other medical reason that the Investigator determines that the subject should not participate in the study
14. Known history of previous pelvic organ prolapse greater than the POP-Q Stage 2 as defined by the international continence society (ICS).

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-08-26 (Actual)

PRIMARY OUTCOMES:
Responder rate at Day 21 | 21 Days
  Responder rate at Day 21, where responder is defined as a subject who has at least 50% reduction in mean 12-hour pad weight test through assessment period of treatment phase (the last 7 days of 14-day device usage period), when compared to the mean pad weight test during the 7-day baseline phase

SECONDARY OUTCOMES:
Percent Change in mean pad weight | 7 Days, 14 Days
  Percent change in mean pad weight during assessment period of treatment phase (the last 7 days of 14-day device usage period), from the mean pad weight during the 7-day baseline phase
Percent change in the frequency of SUI events per the patient diary | 7 Days, 14 Days
  Percent change in the frequency of SUI events per the patient diary, defined as average number of incontinence episodes per 12 hours during assessment period of treatment phase (the last 7 days of 14-day device usage period), from the average of baseline phase
Responder rate for frequency of SUI events per the patient diary at Day 21, | 21 Days
  Where responder is defined as a subject who has at least 50% reduction in the number of incontinence episodes per day during the last 7 days of
Percent change in Incontinence Impact Questionnaire (IIQ-7) score | 21 Days
  7 questions about how urinary incontinence has affected a subjects life. Questions cover physical activity, travel, social relationships and emotional health. The questionnaire asks whether the subjects life has been greatly affected, moderately, slightly or not affected at all.
Percent change in Patient Global Impression of Change (PGIC) score | 21 Days
  It gives a patient reported assessment of change after intervention. The higher the score, the greater the severity (1 being "very much improved"; 7 "very much worse").
Percent change in Incontinence-Quality of Life (I-QOL) Assessment Questionnaire | 21 Days
  The I -QOL consists of 22 items, all of which use a five - point ordinal response scale in which 1 = extremely, 2 = quite a bit, 3 = moderately, 4 = a little, and 5 = not at all. The 22 items can be further grouped into 3 sub-scales: Avoidance and Limiting Behaviour (8 ite ms), Psychosocial Impacts (9 items), and Social Embarrassment (5 items). The total I -QOL and 3 sub scale scores are calculated by summing the unweighted item score and transforming them to a 100 point scale where 0 = mo st severe, and 100 = no problem .
Ease of use per the USE Questionnaire: Usefulness, Satisfaction, and Ease of Use | 21 Days
  The USE questionnaire is meant to be used to assess the Subjective reactions to the usability of the Yōni.Fit ® device. The "Usefulness" section of the questionnaire consists of 19 questions regarding usability of the device scaled from 1- "strongly disagree" to 7- "strongly agree."
Ease of use per the USE Questionnaire: Satisfaction | 21 Days
  The USE questionnaire is meant to be used to assess the Subjective reactions to the usability of the Yōni.Fit ® device. The "Usefulness" section of the questionnaire consists of 7 questions regarding Satisfaction with the device scaled from 1-"strongly disagree" to 7-"Strongly Agree."
Ease of use per the USE Questionnaire:Ease of Use | 21 Days
  The USE questionnaire is meant to be used to assess the Subjective reactions to the usability of the Yōni.Fit ® device. The "Usefulness" section of the questionnaire consists of 11 questions regarding Ease of Use with the device scaled from 1-"strongly disagree" to 7-"Strongly Agree."

CONTACTS AND LOCATIONS:
Overall Officials: Allsion Watkins-Conti, Study Director — Watkins Conti Products. Inc.
Locations (3):
- United States (3):
  - Stanford University School of Medicine, Stanford, California
  - NYU Langone Health, New York, New York
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Escobar C, Sokol ER, Rosenblum N, Milikien D, Echols K. A Randomized Controlled Trial of a Novel Device for Stress Incontinence. Urogynecology (Phila). 2026 Feb 1;32(2):105-115. doi: 10.1097/SPV.0000000000001676. PMID 40288810